CLINICAL TRIAL: NCT04503356
Title: Evaluation of the Effectiveness of the New Surgical Method OMNI in the Treatment of Adult Patients With Open-angle Glaucoma
Brief Title: OMNI in Open-angle Glaucoma Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Iwona Grabska- Liberek, Professor, Centre of Postgraduate Medical Education
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 44/PB/2018
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Open Angle Glaucoma; Cataract; Eye Diseases; Glaucoma
Keywords: glaucoma; open-angle glaucoma; cataract; glaucoma surgery; ophthalmology; OMNI
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract; Eye Diseases; Glaucoma | interventions — Cataract Extraction

STUDY DESIGN:
Intervention Model Description: To prospectively assess the clinical effect of ab-interno transluminal viscodilation and trabeculotomy performed using the OMNI Surgical System as a standalone procedure or in combination with cataract extraction on intraocular pressure (IOP) and the use of ocular hypotensive medications in patients with open-angle glaucoma (OAG).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMNI as a standalone procedure (Active Comparator)
  Interventions: Procedure: OMNI as a standalone procedure
- OMNI combined with cataract surgery (Active Comparator)
  Interventions: Procedure: OMNI combined with cataract surgery

INTERVENTIONS:
Procedure: OMNI as a standalone procedure — It uses a single, self-sealing clear corneal incision with ab-interno transluminal 360 degree viscodilation of Schlemm's canal followed by up to 360 degree trabeculotomy performed using the OMNI Surgical System as a standalone procedure.
  Arms: OMNI as a standalone procedure
Procedure: OMNI combined with cataract surgery — Phacoemulsification with intraocular lens implantation is performed. Then, ab-interno transluminal 360 degree viscodilation of Schlemm's canal followed by up to 360 degree trabeculotomy performed using the OMNI Surgical System.
  Arms: OMNI combined with cataract surgery

SUMMARY:
This single-center, prospective study will assess safety and effectiveness of 360 degree viscodilation followed by up to 360 degree trabeculotomy used in patients with early or moderate open-angle glaucoma in a real-world setting either as a standalone procedure in pseudophakic patients (or phakic) or combined with phacoemulsification cataract procedures.

Medication usage, IOP and secondary surgical procedures necessary for IOP control will be analyzed during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with open-angle glaucoma including pigmentary and pseudoexfoliative glaucoma
* 0-3 topical ocular hypotensive medications at preoperative baseline. Fixed combinations counted as number of components
* Open angles (Shaffer grade ≥3)
* early or moderate glaucoma (based on visual field)
* Subjects with a combined procedure should have had uncomplicated cataract surgery (i.e. intact and centered capsulorrhexis, intact posterior capsular bag, no evidence of zonular dehiscence or rupture, well centered IOL)

Exclusion Criteria:

* Any of the following prior treatments for glaucoma:

  * Suprachoroidal stent
  * Laser trabeculoplasty ≤6 months prior to OMNI procedure
  * Trabecular bypass implanted ≤6 months prior to OMNI procedure
  * Trabeculectomy or other bleb forming procedure including Xen, Express, glaucoma draining device/valve
  * Prior canaloplasty, goniotomy, or trabeculotomy
* Forms of glaucoma other than OAG including: acute angle closure, traumatic, congenital, malignant, uveitic or neovascular glaucoma
* Under treatment with oral carbonic anhydrase inhibitor at the preoperative visit
* Clinically significant ocular pathology, other than age-related cataract and glaucoma. (e.g. wet AMD, uveitis, corneal edema, proliferative diabetic retinopathy, optic neuritis in medical history)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of eyes with a 20% reduction from baseline in IOP at 12 months on the same number, or fewer, ocular hypotensive medications as at the pre-operative baseline | 1 year
Number of Participants wih Postoperative complications | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Iwona Grabska-Liberek, MD, PhD, Principal Investigator — Ophthalmology Clinic Centre of Postgraduate Medical Education, Warsaw, Poland
Locations (1):
- Orlowski Hospital, Centre of Postgraduate Medical Education, Warsaw, Poland